CLINICAL TRIAL: NCT04458571
Title: Effect of CRRT Duration on Solute Removal
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0405
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: AKI; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood samples and Effluent
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The only FDA approved treatment for acute kidney injury(AKI) for patients is Dialysis-also known as renal replacement therapy(RRT). Continuous RRT(CRRT) is the preferred method in the ICU. Patients receiving CRRT with AKI will be recruited to the study where blood and effluent will be collect prior to CRRT initiation and Day 1,2,and 3 following. Metabolites will be assessed to determine solute removal, and also to identify the time at which solute removal has reached steady state. This will help determine the best duration of CRRT.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) occurs in 30-50% of hospitalized patients admitted to the intensive care unit (ICU). Dialysis - also known as renal replacement therapy (RRT) - is the only FDA approved treatment for AKI and continuous RRT (CRRT) is generally the preferred method of RRT in the ICU. The in-hospital mortality of patients with AKI requiring dialysis in the ICU is over 50% which is much greater than other serious illnesses.Unfortunately, the quality of care delivered to patients with AKI receiving CRRT is poor due to practice variability and lack of quality indicators to assess CRRT performance. Since one of the fundamental purposes of CRRT is to remove the build-up of metabolites that accumulate during AKI, accurate methods to assess solute clearance would be especially valuable. Indeed, development of methods to assess solute clearance during CRRT has been identified as a research priority. Although changes in plasma creatinine has been suggested as a potential quality indicator of solute removal during CRRT, no study has assessed how reductions of plasma creatinine over time compare to the reductions of other plasma metabolites. Thus, the duration of CRRT necessary to achieve adequate solute removal is unknown - in fact, there is not yet even an agreed-upon working definition of what adequate solute removal during CRRT should be. The investigators propose to conduct a prospective, single center study of 112 CRRT patients to determine the effect of CRRT duration on solute removal in order to identify the time at which solute removal has reached steady state. To assess solute removal, 102 metabolites will be determined in the plasma and effluent via untargeted ultra high pressure liquid chromatography coupled to mass spectrometry (UHPLC-MS). Metabolites will be assessed on plasma collected immediately prior to CRRT initiation, and on plasma and effluent collected on days 1, 2, and 3 post-CRRT initiation. Steady state is defined as the time point at which a plasma metabolite is not significantly reduced during CRRT - as assessed over a 24 hour time period. Based on preliminary data, the investigators hypothesize that >90% of metabolites will reach steady state by day 2 of CRRT, and that >95% of metabolites will reach steady state by day 3 of CRRT.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients being initiated on CRRT at University of Colorado Hospital (UCH) will be considered for enrollment.

Exclusion Criteria:

* Vulnerable populations such as children, pregnant women, and prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to University of Colorado Hospital and being initiated on CRRT.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Steady State Metabolites | 3 years
  The primary outcome of interest is the binary identification of steady state for each metabolite. Approximately 100 metabolites will be measured including amino acids, phosphorus, creatinine, and BUN

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Faubel, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided